CLINICAL TRIAL: NCT02192346
Title: Phase I Study of Alpha-tocopheryloxyacetic Acid (α-TEA) in Patients With Advanced Cancer
Brief Title: α-TEA in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-043A
Record Dates: First submitted 2014-07-13; First posted 2014-07-16 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Carcinoma; Metastatic Sarcoma; Metastatic Lymphoma
Keywords: metastatic; refractory; progressive
MeSH Terms: conditions — Carcinoma; Sarcoma; Lymphoma; Neoplasm Metastasis | interventions — 2,5,7,8-tetramethyl-2R-(4R,8R,12-trimethyltridecyl)chroman-6-yloxy acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 2.4 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 2.4 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 2.4 mg/kg α-TEA
- 4.8 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 4.8 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 4.8 mg/kg α-TEA
- 8.0 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 8.0 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 8.0 mg/kg α-TEA
- 9.6 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 9.6 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 9.6 mg/kg α-TEA
- 12 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 12 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 12 mg/kg α-TEA
- 16.8 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 16.8 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 16.8 mg/kg α-TEA
- 19.2 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 19.2 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 19.2 mg/kg α-TEA
- 22.3 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 22.3 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 22.3 mg/kg α-TEA
- 26.8 mg/kg α-TEA (Experimental): Patients will receive oral α-TEA 26.8 mg/kg daily for the first 14 days of a 28 day cycle.
  Interventions: Drug: 26.8 mg/kg α-TEA

INTERVENTIONS:
Drug: 2.4 mg/kg α-TEA — Patients receive oral α-TEA 2.4 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 2.4 mg/kg α-TEA
Drug: 4.8 mg/kg α-TEA — Patients will receive oral α-TEA 4.8 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 4.8 mg/kg α-TEA
Drug: 8.0 mg/kg α-TEA — Patients will receive oral α-TEA 8.0 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 8.0 mg/kg α-TEA
Drug: 9.6 mg/kg α-TEA — Patients will receive oral α-TEA 9.6 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 9.6 mg/kg α-TEA
Drug: 12 mg/kg α-TEA — Patients will receive oral α-TEA 12 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 12 mg/kg α-TEA
Drug: 16.8 mg/kg α-TEA — Patients will receive oral α-TEA 16.8 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 16.8 mg/kg α-TEA
Drug: 19.2 mg/kg α-TEA — Patients will receive oral α-TEA 19.2 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 19.2 mg/kg α-TEA
Drug: 22.3 mg/kg α-TEA — Patients will receive oral α-TEA 22.3 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 22.3 mg/kg α-TEA
Drug: 26.8 mg/kg α-TEA — Patients will receive oral α-TEA 26.8 mg/kg daily for the first 14 days of a 28 day cycle.
  Arms: 26.8 mg/kg α-TEA

SUMMARY:
The goal of this study is to find the highest dose of α-TEA that can be given to patients safely, to identify potential side effects of α-TEA, and to measure the amount of α-TEA in patients' blood.

Additional goals of this study are to monitor the effect on tumors, to check for specific immune cells circulating in the blood, and to see if there are certain features of tumors that make it possible to predict the response to α-TEA.

DETAILED DESCRIPTION:
This is a dose-escalation study in which doses ranging from 2.4 mg/kg to 26.8 mg/kg of α-TEA will be tested.

The main clinical objectives of this phase I two-stage dose-escalation trial will be to characterize α-TEA related toxicity, determine the maximum tolerated dose, and pharmacokinetics of α-TEA in humans. Tumor response and exploratory immunological monitoring will also be performed. Specifically, we will determine the frequency of circulating peripheral T cell subset populations including CD4+, CD8+ T cells and their activation status (central memory, effector cells) and regulatory T cells (CD4/CD25/Foxp3). Exploratory monitoring to assess tumor apoptosis and serum cytokine levels will also be performed to gain additional insight on the influence of α-TEA on the immune response and tumor. An assessment of the immunoscore in patients with tumor amenable to biopsy will also provide hypothesis-generating data on the influence of α-TEA on the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable or evaluable metastatic carcinoma, sarcoma or lymphoma who have malignancy refractory or progressed after therapy and for whom no other standard (non-experimental) therapy exists or who have declined available standard therapy, with potential to induce cure, remission or enhanced survival. Either histologic or cytologic diagnosis is acceptable of the primary cancer, or clinical evidence of metastasis.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Age 18 years or above.
* Laboratory values (performed within 28 days prior to enrollment) within protocol specified range.
* Confirmed radiographic and/or serum marker showing cancer progression after at least one systemic therapy for metastatic disease.
* Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand the investigational nature of the study and the risks associated with the therapy.
* No active bleeding.
* No coagulopathy (INR <1.5, PT <16 seconds, PTT < 38 seconds) at baseline.
* Anticipated lifespan greater than 12 weeks.
* Ability to swallow capsules
* Women of childbearing potential must have a negative pregnancy test and must avoid becoming pregnant while on α-TEA and for 4 weeks after the last dose of α-TEA. Men must avoid fathering a child while on α-TEA and for 4 weeks after the last dose of α-TEA.

Exclusion Criteria:

* Active serious infection that could affect treatment.
* Coagulopathy or need for anti-coagulation therapy.
* Malabsorbtion state such as ulcerative colitis, previous surgical resection of > 20% of intestine or stomach.
* History of or active atrial fibrilliationfibrillation or supraventricular tachycardia
* Cardiac ejection fraction less than the lower limit of normal on echocardiography
* Right atrial enlargement on echocardiography
* Active cardiac ischemia. Patients with a history of ischemia ameliorated with stent placement or coronary artery bypass grafting and who have no evidence of ischemia by exercise or physiological stress testing are eligible.
* History of or active congestive heart failure
* Patients with tumor that has invaded vagal nerve, carotid bodies, mediastinal structures, pericardium or myocardium.
* Abnormal thyroid function, or euthyroid, but are on medication for thyroid disorders
* Need for chronic high dose maintenance oral steroids. Stable treatment with prednisone ≤ 10 mg daily (or a biologically-equivalent dose of another steroid) is allowed. Patients who require brief courses of steroids to manage allergic reaction to intravenous contrast used in radiographic studies are eligible. Patients requiring steroids for management of CNS metastatic disease are not eligible.
* Surgery or severe trauma within 4 weeks of study entry (minimally invasive procedures acceptable).
* Active brain metastatic disease. Patients with brain metastases who have been treated with surgery, gamma-knife radiosurgery or radiation and no radiographic progression for at least 4 weeks and off steroids are eligible.
* Any medical or psychiatric condition that in the opinion of the PI would preclude compliance with study procedures.
* Vitamin E supplements
* QTc greater than 450 msec at baseline (calculated using Bazett's formula), sick-sinus syndrome or other active cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 28 Days
  Patients are seen in clinic 7 times over a 28-day period. Patients will have 6 physical exams and meet with a research nurse 5 times for evaluation of any potential drug-related toxicities. In addition, blood will be drawn 7 times for complete blood counts and metabolic panel to check for hematological toxicities. After 28 days, a review of all safety data will determine whether the dose will be increased for subsequent patients.

SECONDARY OUTCOMES:
Number of Adverse Events Possibly Caused by α-TEA | 28 days
  Patients are seen in clinic 7 times over a 28-day period. Patients will have 6 physical exams and meet with a research nurse 5 times for evaluation of any potential drug-related toxicities. In addition, blood will be drawn 7 times for complete blood counts and metabolic panel to check for hematological toxicities. This information will be used to identify toxicities of α-TEA and characterize the safety profile.
Blood serum levels of α-TEA | 28 days
  Patients will have 11 blood draws over 28 days for evaluation of pharmacokinetics. High-performance liquid chromatography (HPLC) and mass spectrometry detection (MSD) will be used to determine serum drug levels of α-TEA using blood samples collected just before the first dose of α-TEA and 1, 4, 8, and 24 hours after the first dose. Additional samples will be drawn just before the α-TEA dose on Days 2, 5, 8, 15, 22, and 29.

OTHER OUTCOMES:
Change in Tumor burden from baseline to 28 days | 28 Days
  Imaging exams (CT, MRI, PET, bone scan, or ultrasound) will be done before treatment and after 28 days to evaluate response to treatment. Imaging modality will be determined by the treating physician.
Change in Activity and Proliferation of Circulating T cell Sub-Populations | 28 days
  Blood will be drawn at before treatment and on days 8 and 29 to identify the type and proportion of circulating T cell subsets.
Change in the Number of Tumor-Infiltrating T cells from Baseline to 35 days | 35 days
  Patients who agree to an optional biopsy and have a subcutaneous or lymph node metastatic site amenable to a simple biopsy procedure will be included in this analysis to evaluate the number of tumor-infiltrating T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Cancer Center, Earle A. Chiles Reserach Institute at the Robert W. Franz Cancer Center
Locations (5):
- United States (5):
  - Providence Oncology & Hematology Care Clinic- Southeast, Clackamas, Oregon
  - Providence Oncology & Hematoloty Care Clinic- Newberg, Newberg, Oregon
  - Providence Oncology & Hematology Care Clinic- Willamette Falls, Oregon City, Oregon
  - Providence Oncology & Hematology Care Clinic- Eastside, Portland, Oregon
  - Providence Oncology & Hematology Care Clinic- Westside, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/